CLINICAL TRIAL: NCT00107939
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy, Safety and Tolerability of Licarbazepine 750 ¿ 2000 mg/d as Adjunctive Therapy to an Atypical Antipsychotic in the Treatment of Manic Episodes of Bipolar I Disorder Over 6 Weeks
Brief Title: Study of Licarbazepine in the Treatment of Manic Episodes of Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLIC477D2302
Record Dates: First submitted 2005-04-11; First posted 2005-04-12 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder; manic episode; treatment; licarbazepine
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — 10,11-dihydro-10-hydroxy-5H-dibenz(b,f)azepine-5-carboxamide

INTERVENTIONS:
Drug: Licarbazepine

SUMMARY:
The purpose of this study is to evaluate the effectiveness and tolerability of an investigational drug for the treatment of manic episodes of bipolar disorder. The investigational drug will be given as additional therapy to one of the five following medications: risperidone, olanzapine, quetiapine, ziprasidone, or aripiprazole. These medications are already FDA (Food and Drug Administration)-approved treatments for mania.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar disorder (type I) with manic or mixed episodes (including patients with/without psychotic features or with/without a history of rapid cycling)
* In need of psychiatric treatment
* Cooperation and willingness to complete all aspects of the study

Exclusion Criteria:

* Current diagnosis other than bipolar I disorder
* History of schizophrenia or schizoaffective disorder
* Drug dependence within 1 month prior to study start or testing positive in a urine drug test
* Suicide attempt within 1 month prior to study start or at immediate risk of harm to self or others
* Any form of psychotherapy within 1 month prior to study start

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2004-11; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Mean reduction in manic episodes and major depressive episodes from baseline to endpoint (week 6)

SECONDARY OUTCOMES:
Safety and tolerability of treatment with licarbazepine over 6 weeks, with respect to adverse events and SAEs, laboratory values, ECGs and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- United States (21):
  - Investigational Site, Little Rock, Arkansas
  - Investigational Site, Orange, California
  - Investigational Site, Pico Rivera, California
  - Investigational Site, San Diego, California
  - Investigational Site, Boca Raton, Florida
  - Investigational Site, Atlanta, Georgia
  - Investigational Site, Chicago, Illinois
  - Investigational Site, Joliet, Illinois
  - Investigational Site, Indianapolis, Indiana
  - Investigational Site, Topeka, Kansas
  - Investigational Site, Kansas City, Missouri
  - Investigational Site, St Louis, Missouri
  - Invetigational Site, Brooklyne, New York
  - Investigational Site, Cedarhurst, New York
  - Investigational Site, New York, New York
  - Investigational Site, Cincinnati, Ohio
  - Investigational Site, Columbus, Ohio
  - Investigational Site, Providence, Rhode Island
  - Investigational Site, Bellaire, Texas
  - Investigational Site, Bellevue, Washington
  - Investigational Site, West Allis, Wisconsin